CLINICAL TRIAL: NCT06343324
Title: The Effect of Web-Based "NIV Living Training" on NIV Compliance and Insomnia Severity in Individuals Using Noninvasive Ventilators (NIV) at Home: Randomized Controlled Study
Brief Title: Effect of Web-Based Adaptation and Insomnia Severity in Individuals Using Noninvasive Ventilators at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Şahabettin Eriş, Nurse, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2023/012
Record Dates: First submitted 2024-03-24; First posted 2024-04-02 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Noninvasive Ventilation; COPD
Keywords: copd; bıpap; cpap; noninvasive ventilation; home type non invasive ventilation; web-based education
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Individuals in the experimental group will be informed about the mobile application. The web-based mobile application called "Training for Living with NIV" prepared by the researcher will be installed on the mobile phone of the individual or his caregiver. They will be asked to log in to the web-based "NIV Living Training" mobile application twice a week to reinforce their knowledge, and text message alerts will be sent via mobile phone. Patient Descriptive Characteristics Form, S³-NIV Questionnaire and Insomnia Severity Index scales will be applied to the experimental group as pre-test data. The scales will be applied again to the experimental group, which continues education for 8 weeks, in the 4th week and the 8th week.
  Interventions: Behavioral: Web-based education
- Control Group (No Intervention): Written educational material was sent to individuals in the control group. Patient Descriptive Characteristics Form, S³-NIV Questionnaire and Insomnia Severity Index scales will be applied as pre-test data to the control group, which is not given any training other than written material. During the 8-week period, the scales will be applied to the control group again in the 4th week and the 8th week. After the 8th week data collection, web-based "NIV Survival Training" will also be given to individuals in the control group.

INTERVENTIONS:
Behavioral: Web-based education — Patients using noninvasive ventilation at home will receive detailed information about accessing, logging in and using web-based training. Pretest data will be collected, then week 4 and week 8 data will be collected.
  Arms: Experimental

SUMMARY:
Home use of the NIV device, which is used to manage respiratory failure, one of the most disturbing symptoms due to COPD, will continue to increase. There is a need for studies evaluating the effectiveness of the use of WEB-based training programs in making patients and their families independent in the use of this device. This study will produce evidence for this effect and contribute to the awareness of healthcare professionals working in this field. The WEB-based training module to be developed aims to increase compliance with NIV in patients using NIV at home for a long time and to manage symptoms such as insomnia that may develop due to NIV.

DETAILED DESCRIPTION:
Support will be received from a software expert in mobile application development. The Mobile Application will be given the short name "Breathe", which indicates that it is an application application. The mobile application is planned to consist of 7 interfaces. 1.Interface: Training on Living with NIV - Password and Information General information about Living with NIV Training will be included. It is an interface where individuals can log in to the system with their password and information.

2.Interface: What is BIPAP? This interface will include general information about individuals' intended use of NIV, what it does, and how to select equipment.

3.Interface: Maintenance and cleaning of the device This interface will contain information on when and how the NIV device and equipment should be cleaned.

4.Interface: Most frequently asked questions about BIPAP treatment This interface will include the problems that individuals frequently experience when using NIV and tips on how to solve these problems.

Interface 5: Insomnia and coping methods This interface will contain information about insomnia and what techniques to use to cope with insomnia. It will also include sleep exercise to help you fall asleep.

6.Interface: Trainings This interface; It will consist of educational content such as breathing exercise, lung cleaning technique, breathing control in daily life activities (walking, bathing, climbing stairs, etc.), personal hygiene and dressing, and communication and special situations while using NIV.

7.Interface: Communication It is an interface where individuals can communicate with the researcher and ask questions.

Individuals assigned to the experimental group Individuals in the experimental group will be informed about the mobile application. The web-based mobile application called "Training for Living with NIV" prepared by the researcher will be installed on the mobile phone of the individual or his caregiver. They will be asked to log in to the web-based "NIV Living Training" mobile application once a week to consolidate their knowledge, and text message alerts will be sent via mobile phone. S³-NIV Questionnaire and ISI forms will be applied to the experimental group again in the first week, 4th week and 8th week.

Individuals assigned to the control group Written educational material was sent to individuals in the control group. S³-NIV Questionnaire and ISI forms will be applied again to the control group in the first week, 4th week and 8th week. After the 8th week data collection, web-based "NIV Survival Training" will also be given to individuals in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have used NIV at home for at least 4 months or more,
* Individuals between the ages of 50-75,
* No communication barrier,
* Whether the caregiver or the individual himself is using a smart phone,
* Having internet access,
* Ability to read and understand Turkish.

Exclusion Criteria:

* Myocardial infarction or cerebrovascular accident, schizophrenia, etc. in the last 3 months. Individuals who cannot provide their own self-care due to illness,
* Being diagnosed with cancer,
* Being hospitalized with acute exacerbation,

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Patient Identifiable Characteristics Form | 1 minute
  This form, prepared by the researcher using the literature, consists of 8 questions regarding the patients' sociodemographic (age, gender, education, etc.) and clinical characteristics (disease type, etc.).

SECONDARY OUTCOMES:
S³-NIV Questionnaire | 3 minute
  The questionnaire was developed to evaluate noninvasive ventilation at home. The survey consists of 10 items and two sub-dimensions. A five-point Likert scale is used to rate the items: always yes (0), mostly yes (1), sometimes yes (2), mostly no (3), completely no (4). The Cronbach alpha reliability coefficient of the survey was found to be 0.77.
  Score of the survey total and sub-dimensions; It is obtained by taking the average of the total score of the items and multiplying the result by 2.5. The lowest possible score (0) corresponds to the highest impact of disease and treatment, while the highest possible score (10) corresponds to the lowest impact of disease and treatment.

OTHER OUTCOMES:
insomnia severity index | 5 minute
  This scale, developed to determine the severity of insomnia, is used in normal population screening and clinical evaluation of insomnia. 7 items and two subscales It is a 5-point Likert type scale. Each item is scored between 0 and 4, and the total score varies between 0-28 points. Scores of 0-7 on the scale indicate clinically insignificant insomnia, 8-14 indicates mild insomnia, 15-21 indicates moderate insomnia, and 22-28 indicates severe insomnia.
  The internal consistency coefficient of the scale was found to be 0.79.
Expected behavioral changes in the individual survey | 1 minute
  It was developed by the researcher to evaluate 6 behaviors that are expected to change and develop in individuals in 8 weeks as a result of web-based training.

CONTACTS AND LOCATIONS:
Overall Officials: Şahabettin ERİŞ, MScN, Principal Investigator — study principal investigator
Locations (1):
- Health Sciences University Konya Beyhekim Training and Research Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data will be collected by the researcher at the University of Health Sciences Konya Beyhekim Training and Research Hospital.